CLINICAL TRIAL: NCT03377192
Title: Impedance Pneumography in Assessment of Asthma Control in Preschool Children
Acronym: IPAAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: HUS Skin and Allergy Hospital (Other)
Collaborators: Revenio Research (Industry); Mehiläinen (Unknown)
Responsible Party: Principal Investigator, Pekka Malmberg, MD, PhD, Head of clinical physiology, HUS Skin and Allergy Hospital
Other Study IDs: VCS-002
Record Dates: First submitted 2017-12-05; First posted 2017-12-19 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Wheezing; Asthma in Children
Keywords: Impedance pneumography; Respiratory function; Asthma management
MeSH Terms: conditions — Respiratory Sounds; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the value of impedance pneumography, used as overnight home recordings during a longitudinal design, in assessing asthma control in preschool children

DETAILED DESCRIPTION:
Lung function assessment of preschool children is hindered by their limited co-operation in conventional tests such as peak expiratory flow (PEF) or spirometry. However, indices derived from spontaneous tidal respiratory air flow and the shape of tidal expiratory flow-volume and flow-time curves relate to lung function and are easier to record even in young children. As a more advanced approach, the time dynamics and complexity properties of the tidal breathing flow volume (TBFV) signal have been analysed and found to relate to various respiratory conditions.

Impedance pneumography (IP) is a method for measuring changes in the thoracic electrical impedance through skin electrodes, which varies as a function of lung aeration i.e. breathing. Recent technical advancements have enabled IP to be used for accurate non-invasive tidal flow signal measurement. Moreover, in overnight recordings at home, IP was found feasible for quantifying nocturnal TBFV variability in young children with lower respiratory symptoms, showing that preschool children with high risk of asthma present with increased variation of tidal flow profile shape, and momentarily lowered chaoticity, compared to children with lower risk of asthma. So far, there are no studies that have addressed the utility of IP to assess asthma control in young children with asthma.

The purpose of this study is to investigate the utility of a commercially available IP device (VENTICA, Icare Finland, Finland) and IP-derived clinical indices in assessing the clinical control of asthmatic children receiving normal therapy in a longitudinal setting. The primary hypothesis is that TBFV variability quantified by IP is associated with disease control during management of young children with asthma. The secondary hypothesis is that TBFV variability quantified by IP predicts changes in disease control during management of young children with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-7 years, both sexes
* Attending pediatric ward in the study centre due to asthmatic symptoms (wheeze, cough and/or dyspnea)
* History and clinical signs allowing diagnosis of doctor diagnosed asthma and the need to start regular anti-asthmatic medication
* Signed informed consent

Exclusion Criteria:

* Use of inhaled corticosteroid medication 30 days prior to study entry
* Other cardiorespiratory or neurological chronic diseases or states that may affect breathing
* Acute respiratory infection 2 weeks prior to study entry
* Chronic respiratory disorder of prematurity
* Implanted or external active medical devices

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Thirty (30) patients who have attended pediatric ward in the study centre(s) due to asthmatic symptoms (wheeze, cough, dyspnea) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Childhood asthma control test (C-ACT) | Weekly up to maximum 6 months or until loss of asthma control/exacerbation
  Questionnaire that measures current asthma control, including 7 questions and a minimum score of 0 and maximum score of 27; score 19 or less indicates that asthma is not controlled.

SECONDARY OUTCOMES:
Time-to-response (TTR) | Minimum of 30 days from initiation of anti-asthmatic medication up to max 6 months
  Duration from visit 1 to good asthma control (C-ACT>19)
Time-to-loss-of-control (TTLOC) | Minimum of 30 days from initiation of anti-asthmatic medication up to max 6 months
  Duration from the visit 2 and 3 until loss of asthma control (C-ACT<16) or asthma exacerbation
Lung function | Every visit up to maximum 6 months
  Respiratory resistance and exercise induced increase in resistance, measured by the oscillometric method

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Malmberg, MD, PhD, Principal Investigator — HUS Skin and Allergy Hospital
Locations (2):
- Finland (2):
  - HUS Skin and Allergy Hospital, Helsinki
  - Mehiläinen Paediatric Allergy Clinic, Helsinki

REFERENCES:
- [Derived] Burman J, Malmberg LP, Remes S, Jartti T, Pelkonen AS, Makela MJ. Impulse oscillometry and free-running tests for diagnosing asthma and monitoring lung function in young children. Ann Allergy Asthma Immunol. 2021 Sep;127(3):326-333. doi: 10.1016/j.anai.2021.03.030. Epub 2021 Apr 2. PMID 33819614